CLINICAL TRIAL: NCT04575207
Title: A Prospective, Multicenter, Blinded, Randomized, Noninferiority Clinical Trial of Coronary Angiography Fractional Flow Reserve (caFFR) Versus Fractional Flow Reserve (FFR) to Guide Percutaneous Coronary Intervention（Flash FFR Ⅱ ）
Brief Title: The Flash FFR Ⅱ Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Rainmed Ltd., Suzhou, China (Unknown)
Responsible Party: Principal Investigator, Yong Huo, Chief physician of cardiology Department, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SZRMD2020001
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Myocardial Ischaemia; Coronary Circulation; Stable Angina Pectoris; Unstable Angina Pectoris; Asymptomatic Ischemia; Acute Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: Flash; FFR; caFFR; coronary angiography-derived fractional flow reserve; Coronary Artery Disease; Myocardial Ischaemia; Percutaneous Coronary Intervention; Coronary Circulation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Angina, Stable; Angina, Unstable; photopsia | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the Flash FFR II study, clinical outcome assessors (including the follow-up research personnel, clinical events committee (CEC), data and safety monitoring board (DSMB), and core laboratory) will be blinded to randomization arm. The data safety monitoring board (DSMB) may request unblinding of grouping information due to patient safety reasons. All the study site personnel will receive training for the blinding requirements before the trial initiating to prevent disclosure of random assignment to the follow-up personnel in any unplanned way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caFFR-guided (Experimental): Participants who are randomly assigned to caFFR-guided group will receive the detection of Coronary Angiography-Derived Fractional Flow Reserve (caFFR) Measurement System. The online caFFR value is used to guide the PCI strategy. If caFFR ≤ 0.80, PCI treatment will be performed in lesions and optimal medicine treatment will be performed when caFFR > 0.80.
  Interventions: Diagnostic Test: caFFR
- FFR-guided (Active Comparator): Participants who are randomly assigned to FFR-guided group will receive the detection of pressure wire. The FFR value is used to guide the PCI strategy. If FFR ≤ 0.80, PCI treatment will be performed in lesions and optimal medicine treatment will be performed when FFR > 0.80.
  Interventions: Diagnostic Test: FFR

INTERVENTIONS:
Diagnostic Test: caFFR — caFFR is a new index of physiological assessment of coronary artery stenosis severity, based on angiographic images. Through two-dimensional analysis and three-dimensional reconstruction of two coronary angiography image series with an angle-off > 30 degrees, combined with fluid mechanics, TIMI frame counting method, and optimized CFD algorithm, the pressure drop from coronary ostium to every point in the vessel can be obtained, and then the caFFR value of each point in the vessel can be computed. The cutoff value in this trial is caFFR ≤ 0.80 for myocardial ischemia.
  Other Names: Coronary Angiography-Derived Fractional Flow Reserve
  Arms: caFFR-guided
Diagnostic Test: FFR — FFR is a widely used, pressure-based functional assessment index of coronary stenoses obtained with an intracoronary pressure wire fitted with pressure sensors. The pressure wire passes through the stenosis and directly measures the pressure distal to the stenosis. FFR value can be obtained by combining the pressure at the coronary ostium and the distal pressure to the stenosis. The cutoff value in this trial is FFR ≤ 0.80 for myocardial ischemia.
  Other Names: Fractional Flow Reserve
  Arms: FFR-guided

SUMMARY:
The overall purpose of Flash FFR Ⅱ is to investigate whether coronary angiography-derived fractional flow reserve (caFFR), compared with fractional flow reserve (FFR) measured by a pressure wire, has non-inferior clinical effect and cost benefit in guiding the percutaneous coronary intervention (PCI) for patients with moderate coronary artery stenosis in terms of long-term clinical prognosis.

DETAILED DESCRIPTION:
Flash FFR Ⅱ is a prospective, multicenter, blinded, randomized, non-inferiority trial. Eligible patients with moderate coronary artery stenosis will be included in the study and randomly assigned to either caFFR-guided group or FFR-guided group. Participant caFFR or FFR will be used to guide percutaneous coronary intervention (PCI) strategy.

The rate of major cardiovascular adverse events (MACE) and the cost data will be collected during the long-term follow-up (2 years). MACE is defined as a composite of all-cause death, myocardial infarction (MI), unplanned revascularization. Clinical outcomes and cost-effectiveness will be compared between the two groups.

A subgroup analysis is pre-set and included in the protocol, including age, sex, body mass index, diabetes mellitus, smoking status, mean aortic pressure (resting state), acute coronary syndrome, left ventricular ejection fraction, lesion site, lesion stenosis severity, target vessel reference diameter, small vessel lesion, blood flow velocity, PCI mode, and so on.

The trial is equipped with a core laboratory. Some interesting sub-studies will be carried out, such as a comparison of laboratory and operator analysis results.

If the trial results show non-inferiority, it should be noted that caFFR can bring new benefits to both operators and patients as a new index of physiological assessment of coronary artery stenosis severity with the advantages of lower cost, less risk, faster time, and less use of resources.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  1. Age above 18 years old, no limit on the gender;
  2. Angiography is considered necessary and feasible by investigator, and PCI will be performed if necessary;
  3. Suspected coronary heart disease, stable angina pectoris, unstable angina pectoris, non-culprit vascular assessment in participants with acute non-ST-segment elevation myocardial infarction, and non-culprit vascular assessment in patients with previous ST-segment elevation acute myocardial infarction;
  4. Participants voluntarily participate in this clinical trial and sign informed consent form.
* Coronary angiography inclusion criteria:

The presence of at least one stenosis and meets the following imaging findings:

1. The degree of coronary artery stenosis≥50% and ≤90% by visual measurement;
2. The reference diameter of the stenotic segment≥2.25 mm by visual measurement;
3. The investigator visually observes the target vessel through angiographic images, and consider that PCI surgery is technically feasible.

Exclusion Criteria:

* General exclusion criteria:

  1. Acute ST-segment elevation myocardial infarction within 6 days;
  2. Cardiogenic shock or left ventricular ejection fraction≤50%;
  3. eGFR < 30 mL/min (1.73 m2);
  4. Severe coagulation dysfunctions or bleeding disorders;
  5. Allergic to iodine contrast medium or contraindications for adenosine administration;
  6. Severe aortic stenosis;
  7. Life expectancy less than 1 year;
  8. Pregnant women or women planning a recent pregnancy;
  9. Participation in any other clinical trials of devices or drugs (ongoing or within the past 1 month);
  10. The investigator believes that the particitant has other conditions that are not suitable for clinical trials.
* Coronary angiography exclusion criteria:

  1. TIMI flow in the target vessel<grade III ;
  2. Presence of myocardial bridge and systolic compression ≥50% in the target vessel;
  3. Presence of artificial bypass in the target vessel;
  4. Left main coronary artery or right coronary artery ostial lesions;
  5. Stent implantation in the target vessel within 3 months;
  6. Target vessel provides collateral support to chronically total occluded vessels;
  7. Presence of factors affecting angiographic analysis and stenosis visualization, including incomplete vessel opacification, or overlap with other coronary branches of extreme vessel foreshortening.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2132 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year
  A composite of all-cause death, myocardial infarction (MI), and unplanned revascularization

SECONDARY OUTCOMES:
MACE（excluding PCI-related MI） | 1 month, 1 year, 2 years
  A composite of all-cause death, myocardial infarction (excluding PCI-related), and unplanned revascularization
Death | 1 month, 6 months, 1 year, 2 years
  Cardiovascular, non-cardiovascular, and undetermined death
MI | 1 month, 6 months, 1 year, 2 years
  Target vessel related and non-target vessel related MI
Target vessel revascularization (TVR) | 1 month, 6 months, 1 year, 2 years
  The ischemia driven and non-ischemia driven TVR
Any coronary artery revascularization | 1 month, 6 months, 1 year, 2 years
  The ischemia driven and non-ischemia driven revascularization
Definite or probable stent thrombosis | 1 month, 6 months, 1 year, 2 years
  Definite and probable stent thrombosis during acute, sub-acute, late, and very late phase
Evaluation of health economics | 1 month, 6 months, 1 year
  Cost-utility analysis and computation of incremental cost-effectiveness ratio.
Analysis of participant discomfort during the operation (none/mild/moderate/severe ) | During the operation
  During the caFFR or FFR detection, the operator will ask the participant if there is discomfort (none/mild/moderate/severe ) and what kind of discomfort(such as palpitation, chest stuffy , nausea, dizziness, foreign body invasion ), and fill out a questionnaire after the operation.The discomfort of all participants caused by the use of drugs, intervention, etc. during the caFFR or FFR detection will be analyzed.
The changes of PCI strategy depending on caFFR/FFR information | During the operation
  Before randomization,the operators will be asked to provide their planned treatment strategy based on the angiographic information alone.
  After randomization and functional assessment,we will record how caFFR/FFR changed the treatment strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, MD, Study Chair — Peking University First Hospital
Locations (13):
- China (13):
  - Beijing Hospital of Traditional Chinese Medicine, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The University of Hong Kong Shenzhen hospital, Shenzhen, Guangdong
  - The People's Hospital of Hebi, Hebi, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - QILU Hospital of Shandong University, Jinan, Shandong
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - Department of Cardiology, Peking University First Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Gong Y, Wang W, Yang Q, Liu B, Lu Y, Xu Y, Huo Y, Yi T, Liu J, Li Y, Xu S, Zhao L, Ali ZA, Huo Y. Accuracy of computational pressure-fluid dynamics applied to coronary angiography to derive fractional flow reserve: FLASH FFR. Cardiovasc Res. 2020 Jun 1;116(7):1349-1356. doi: 10.1093/cvr/cvz289. PMID 31693092
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438